CLINICAL TRIAL: NCT03655769
Title: Functional Magnetic Resonance Imaging (fMRI) Analysis of Aging and Awareness in Conditioning
Brief Title: fMRI Analysis of Aging and Awareness in Conditioning
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NA_00045404; R01AG021501 (NIH)
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Transcranial Direct Current Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham tDCS (Sham Comparator): tDCS delivered for only 30 sec to replicate tingling sensation and blind subject
  Interventions: Device: sham transcranial direct current stimulation
- cathodal tDCS (Experimental): cathodal tDCS, 2 milliamps (mA), delivered to right parietal region
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — transcranial direct current stimulation applied at 2 mA over the right parietal region for 20 min
  Arms: cathodal tDCS
Device: sham transcranial direct current stimulation — transcranial direct current stimulation applied at 2 mA over the right parietal region for 30 sec
  Arms: sham tDCS

SUMMARY:
Cathodal Transcranial direct current stimulation (tDCS) was administered to the right parietal region in order to determine if this stimulation could disrupt awareness of the conditioned stimulus (CS) - unconditioned stimulus (US) relationship in a classical conditioning experiment.

ELIGIBILITY:
Inclusion Criteria:

* Educational attainment of at least eight years and English as the native language
* Mini-Mental State Examination (MMSE) score of 26
* Normal episodic memory (i.e., CERAD word List Recall > 5)
* Informed consent; 5) age of 20-30

Exclusion Criteria:

* Disturbed consciousness
* Other neurological or systemic disorder which can cause dementia or cognitive dysfunction
* Prior history of a major psychiatric disorder
* History of definite stroke
* Focal lesion on MRI exam
* Use of anxiolytic, antidepressant, neuroleptic, or sedative medication
* Predominately left-handed
* Has MRI contraindication such as pacemaker, implanted pumps, shrapnel, etc. (full MRI screening form will be filled out).

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-11-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CS-US Awareness | recorded immediately after the 20 minutes of tDCS stimulation
  To assess CS-US awareness, we used a questionnaire The questionnaire consists of 7 true/false questions about the sequence and co-occurrence of the conditioned stimulus (CS, a 1000 Hz tone) and unconditioned stimulus (US, a 100 ms puff of air to the eye). The score can thus range from 0 to 7. Higher score values indicate better awareness of the sequence and co-occurrence of the CS and US

SECONDARY OUTCOMES:
Line bisection test of left-hemifield neglect | recorded immediately after primary awareness questionnaire
  The subject is given a sheet of paper with a number of horizontal lines on it. The subject is instructed to cut each line in half by drawing a small pencil mark through each line. The test is scored by measuring the percent deviation, which is calculated by the following formula:
  Percent deviation=100 x (measured left half - true half)/true half This yields positive numbers for marks placed to the right of center, and negative numbers for marks placed to the left of center. Patients with right hemisphere damage and contralateral neglect show higher positive line bisection scores compared to healthy controls or patients without right hemisphere damage and vice versa.
Eyeblink conditioned responding | recorded during the tDCS administration
  Eyeblink conditioning is recorded while the subject watches a silent movie. For conditioning, the conditioned stimulus (CS) is a 1350 ms 1000 Hz tone. This tone co-terminates with a 100 ms left corneal airpuff (5 psi). 30 CS-US presentations are delivered at an average rate of one every 18 sec. Conditioned responses (CRs) are defined as follows: the difference between the maximum and minimum responses in a 500 ms pre-US time window must exceed four times the standard deviation of the mean of the baseline period (250 ms pre-CS presentation). The 500 ms pre-US time window was selected to minimize the inclusion of voluntary and alpha responses as CRs. Performance is expressed as % CRs, that is, the percent of trials in which a CR occurred. Greater numbers indicate greater amounts of learning.

CONTACTS AND LOCATIONS:
Overall Officials: John Desmond, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No